CLINICAL TRIAL: NCT00410865
Title: Clinical Protocol for Wild Type p53 Gene Induction in Premalignancies of Squamous Epithelium of the Oral Cavity and Oral Pharynx Via an Adenoviral Vector [NCI Supplied Agent Ad-p53, (INGN 201) (Advexin®) NSC 683550, IND# 7135]
Brief Title: Wild Type p53 Adenovirus for Oral Premalignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor withdrawl prior to study completion.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-193
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Mouth Cancer
Keywords: Oral Premalignancies; Mouth Cancer; Dysplasia/Carcinoma in Situ (CIS) of the Oral Cavity; Dysplasia/Carcinoma in situ (CIS) of the Oral Pharynx; Advexin; Gene Therapy; INGN 201; Wild Type p53 Gene Induction
MeSH Terms: conditions — Mouth Neoplasms; Carcinoma in Situ | interventions — advexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- INGN 201 (Experimental): INGN201 injection + oral rinse, day 1, courses 1-6. Twice-daily oral rinses, days 2-5, courses 1-6.
  Interventions: Genetic: INGN 201

INTERVENTIONS:
Genetic: INGN 201 — Mouth rinse given one time on the first day and two times on Days 2-5 of each course of INGN 201. The injection and rinse (first day of each cycle), or the two rinses (Days 2-5 of each cycle), will be separated by at least two hours.
  Other Names: Advexin; Ad-p53

SUMMARY:
Primary Objectives:

1. To determine the maximum tolerated dose and transduction efficiency of adenoviral mediated wild type p53 gene transfer in premalignancies of the upper aerodigestive tract.
2. To determine the efficacy of single agent adenoviral mediated wild type p53 gene transfer in reversing oral premalignancies.

DETAILED DESCRIPTION:
Some cancers that occur in the mouth may in some way be due to a defect in a gene called the p53 gene. In this study, an adenovirus is used as a tool (a "vector") to deliver the normal p53 gene into cells. The parts of the adenovirus that allow it to reproduce and promote infection are removed, and the experimental gene (p53) is added.

Prior to beginning this study, all participants will have a complete medical history and physical exam, including measurement of vital signs and weight. Participants will have an electrocardiogram (ECG), a urine test, and blood tests, including an HIV test. At mid-cycle, another white blood cell count will have to be drawn. Women able to have children must have a negative blood pregnancy test. Participants will be asked what medications have been taken in the past 30 days. Additionally, a chest x-ray will be performed.

All participants will undergo a complete head and neck examination. This includes both visual [direct as well as mirror (and fiberoptic if required)] of all mucosal sites from the nasal and lip areas to the back of the throat. The physician will manually examine areas of the skin, salivary glands, the neck, and thyroid bed. Also, the doctor will make sure the cranial nerves are working properly. Location and size of lesion(s) will be recorded and measured in two dimensions. All lesions present will be photographed prior to the start of the intervention.

Physical examination including a fiberoptic exam, is the established standard of evaluating pre-cancerous lesion(s). Only if a concern for cancer is present , or symptoms are beyond those findings of the physical examination will a CT or MRI be prescribed. These tests (CT and MRI) should not have to be done since they have no established role in the evaluation, management, or follow-up of these lesion(s). If utilized, a CT (computerized tomography) scan is a special test using x-ray along with a computer to give detailed pictures of parts of the body. An MRI (magnetic resonance imaging) is a special test using a strong magnetic field and radio frequency signals to give detailed pictures of parts of the body. An x-ray shows a 2-dimensional picture while a CT scan or an MRI shows 3 dimensions.

Each study course includes one week of treatment followed by three weeks of observation. The length of the study is 6 months (6 courses) for most participants. Participants will return to the clinic twice a day for Days 2 - 5 for each month of participation, and should expect to spend a total of about 6 hours a day at the clinic.

Participants in this study will receive INGN 201 in two ways. The first way will be by injection in the area of the lesion. The second way will be by mouth rinse. Vital signs will be checked each time before participants receive INGN 201. The injection will be given on the first day of each week of the course, after a numbing (anesthetic) medication is applied to prevent discomfort.

The mouth rinse will be given one time on the first day and two times on Days 2 - 5 of each course of INGN 201. The injection and rinse (first day of each cycle), or the two rinses (Days 2 - 5 of each cycle), will be separated by at least two hours. There will be a 30 second rinse with 5% acetic acid, a raspberry flavored, vinegar-like liquid, followed by a tap water rinse just before participants receive INGN 201. Participants will be asked to hold the INGN 201 in their mouth for 30 minutes. Eating and drinking should be avoided for one hour after receiving the mouth rinse. The injection and rinse series will be repeated on a monthly basis for a period of six months.

Participants will be requested to have two biopsies (small tissue samples) of the premalignant lesion taken on Day 5 of the 1st and 6th courses. These biopsies will contribute to the understanding of how the experimental agent works on pre-cancerous cells. In particular, the biopsies will help to determine if the experimental agent is effective in killing pre-cancerous cells (this process is called apoptosis). These studies will also determine if the gene therapy injections have been effective in delivering the gene (p53) to the precancerous cells.

Participants will be observed for three more weeks after the sixth course of treatment. At the end of the study, 28 days after the last dose of INGN 201, participants will have a physical exam, including measurement of weight and vital signs. Participants will have a medical history and blood and urine tests. These tests are done to monitor the effects of the study treatment.

Participants who develop severe side effects will be taken off study, though they may continue to receive follow-up evaluations to monitor their health. Participants will be counseled by their physician should the lesion(s) progress to cancer during the study or follow up period. After counseling, participant may choose to have surgery to remove the precancerous lesion(s), laser surgery, or observation. The participant will then be monitored closely.

Study participants will be followed for five years, and must agree to stay in contact with their personal doctor or the doctor responsible for this study even if they move after the study ends. The participant's personal doctor may be asked to provide information about any anticancer treatments received after the study's completion, as well as information about the patient's overall health.

This is an investigational study. This experimental use of human genes is an example of gene therapy. This is the first time that adenovirus gene therapy has been used for a pre-cancerous condition. This is the first study to use INGN 201 as a mouth rinse. A total of 20 patients will be enrolled at M. D. Anderson. A maximum of 51 subjects will be entered in this multi-center study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged 18 years and older.
* Patients must have histologically confirmed diagnosis of mild-moderate dysplasia or severe dysplasia/carcinoma in situ (CIS) of the oral cavity or oral pharynx.
* Patients must have clinical evidence of mild to moderate dysplasia or severe dysplasia/CIS of the oral cavity or oral pharynx that is diffuse.
* Patients must have diffuse* premalignant disease of the oral cavity or oral pharynx and must have: a) been previously treated with conventional treatment (e.g.: radiation or surgery) for a prior head & neck malignancy or b) failed biochemoprevention approaches for premalignant disease or c) failed other therapeutic approaches for premalignant disease. (*See protocol for definition of diffuse.)
* All patients must have a Karnofsky performance status of greater than or equal to 70% (Karnofsky scale, Appendix B).
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the institution.
* If female and of childbearing potential (non-childbearing defined as 1 year post menopause or surgically sterilized), patients must have a negative serum pregnancy test. Patients (male and female) must agree to use barrier contraception while on study and to avoid pregnancy for 1 year after treatment.
* Patients must have negative serology for the Human Immunodeficiency Virus (HIV) Type I. (Safety of the product has not been established or studied in immunosuppressed populations).
* Patients must have adequate bone marrow function (defined as peripheral absolute granulocyte count of greater than or equal to 2,000/ul and platelet count of greater than or equal to 100,000/ul), adequate liver function (bilirubin less than or equal to 1.0 mg/dl), and adequate renal function (creatinine less than or equal to 1.5 mg/dl).
* Patients must not knowingly be in contact with former tissue or organ transplant recipients and persons known to them to be suffering from severe immunodeficiency disease (either acquired or congenital) during treatment or within 28 days following the last dosing with Ad5CMV p53 (INGN 201).

Exclusion Criteria:

* Active squamous cell carcinoma of the head and neck.
* History of prior malignancies (excluding non-melanoma skin cancers and aerodigestive cancers) unless curatively treated and disease free for greater than or equal to 2 years.
* Prior experimental therapy oral, systemic, topical, or directly injected into the lesion selected for treatment in this study, or radiation directly involving the lesion selected in the last three (3) months.
* Chemotherapy within 21 days prior to study (42 days for mitomycin C and nitrosoureas).
* Pregnant or lactating females. (Transplacental transfer and excretion in breast milk have not been studied with this agent).
* Active systemic viral, bacterial, or fungal infections requiring treatment.
* Patients with serious concurrent illness of psychological, familial, sociological, geographical or other concomitant conditions which do not allow for adequate follow up and compliance with the study protocol.
* Concurrent use of other investigational agents.
* Prior use of any other investigational agent requires a washout period of 8 weeks.
* Any immunosuppressive therapy (including corticosteroids > 10 mg/day) of prednisone or the equivalent.
* Aspirin use in an average dose of >175 mg/d.
* Patients evaluated by Internal Medicine with a baseline blood pressure of > or equal to 140/90 and deemed hypertensive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-06; Primary Completion 2008-03 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of INGN 201 | Following 1 week of experimental treatment in each 4 week course
  MTD is defined as the highest dose level at which there are less than or equal to 1/6 patients with a dose limiting toxicity (DLT).

CONTACTS AND LOCATIONS:
Overall Officials: Gary L. Clayman, MD, Principal Investigator — U.T. MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org